CLINICAL TRIAL: NCT01412580
Title: The Contribution of Health in Utero to Capacity Formation, Education and Economic Outcomes: Experimental Evidence From Tanzania
Brief Title: In Utero Capacity Formation and Socio-economic Outcomes
Acronym: CDS
Status: Completed | Type: Observational
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Plamen Nikolov, Study Director, Harvard University
Other Study IDs: F19899-101
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Folic Acid Deficiency
MeSH Terms: conditions — Folic Acid Deficiency

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- observational followup: This was an observational follow-up to a larger study in which treatment group was given 20 mg of vitamin B1, 20 mg of vitamin B2, 25 mg of vitamin B6, 100 mg of niacin, 50 μg of vitamin B12, 500 mg of vitamin C, 30 mg of vitamin E, and 0.8 mg of folic acid
  Interventions: Other: observational follow-up

INTERVENTIONS:
Other: observational follow-up — observational follow-up

SUMMARY:
Because of the high returns of schooling in developing countries, policymakers pay a lot of attention to increasing school access. But if the mother is deficient in key micronutrients, brain development can biologically constrain children's demand for education. To execute this strategy, the investigators collect cohort observational data on a previous randomized controlled trial with micronutrient supplements offered to HIV-negative pregnant women in Dar es Salaam, Tanzania, between 2001 to 2003.

DETAILED DESCRIPTION:
This is a cohort study which collected follow-up observational data on households which were offered micronutrient supplements. The followup study outcomes include various socio-economic household characteristics and parental post-natal behaviors.

ELIGIBILITY:
These were individuals from the larger study and this study is an observational follow-up.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals from a larger study and this study is an observational follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2002-04; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Children's Cognitive Development | During 2011-2012 (1 year)
Children's Health | During 2011-2012 (1 year)
  BMI, Disease Incidence, Self-reported health
Parental Postnatal Investment Behavior | During 2011-2012 (1 year)
  Outcomes on parental care: care, cognitive stimulation, within-household time and money allocation
Educational Status | During 2011-2012 (1 year)
  School attendance, Student performance (at school), Test Performance

SECONDARY OUTCOMES:
Parental Labor Force Participation | During 2011-2012 (1 year)
  Parent's labor force outcomes: labor status, wages, type of job

CONTACTS AND LOCATIONS:
Overall Officials: Plamen Nikolov, Study Director — Harvard University
Locations (1):
- MUHAS, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No